CLINICAL TRIAL: NCT07229131
Title: Effect of an Oral Acerola Juice Powder on Skin Beauty Parameters in Women Exposed to Environmental Stresses: A Double-blind, Randomised, Placebo-controlled Study.
Brief Title: Effect of an Oral Acerola Juice Powder on Skin Beauty Parameters in Women Exposed to Environmental Stresses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diana SAS (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Organization: Symrise Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GZ25205020P
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pollution; Exposure
Keywords: Skin; Beauty; Environmental stress; Acerola; Vitamin C; Polyphenols

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acerola Juice Powder 1200 mg/day (Experimental): Higher dose
  Interventions: Dietary Supplement: Acerola Juice Powder 1200 mg/day
- Acerola Juice Powder 600 mg/day (Experimental): Lower dose
  Interventions: Dietary Supplement: Acerola Juice Powder 600 mg/day
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Acerola Juice Powder 1200 mg/day — 4 capsules per day, each capsule containing 300mg of Acerola and 100 mg of maltodextrin
  Arms: Acerola Juice Powder 1200 mg/day
Dietary Supplement: Acerola Juice Powder 600 mg/day — 4 capsules/day, each capsule containing 150 mg of Acerola and 250 mg of Maltodextrin
  Arms: Acerola Juice Powder 600 mg/day
Other: Placebo — 4 capsules per day, each capsule containing 400 mg of maltodextrin
  Arms: Placebo

SUMMARY:
The study is being conducted to evaluate the efficacy and the safety of an oral acerola-based product on skin ageing parameters.

DETAILED DESCRIPTION:
The main objective of this study is to assess efficacy of the product on skin translucency after 84 days of product compared to a placebo. The study will also evaluate the effect of the product on different skin parameters (radiance, firmness, elasticity, skin barrier function, skin pH, blood flow) with different instruments. The quality of life and the improvement of skin properties will also be collected with questionnaires completed by the subjects. Finally, the safety of this product will be assessed by collecting all adverse events that might occur during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women.
2. Chinese.
3. Age: in each group of products

   * 50% of subject having 30 to 45 years old
   * 50% of subject having 46 to 60 years old
4. Phototype: II to IV.
5. Subject with dull skin from grade 3 to 7 on skin dullness 9 points scale.
6. Subject exposed to high air pollution up to 2 to 3 hours per day (traffic roads, cigarette smoke, dusts or small particles).
7. Subject who accepts daily exposition to blue light (mobile phone, Ipad, laptop or get exposure to LED light) at home (at least 2h).
8. Subject with at least 1 spot on the face.
9. Subject with BMI ≤ 30
10. Subject, psychologically able to understand the study related information and to give a written informed consent.
11. Subject having given freely and expressly her informed consent.
12. Subject agreeing to not change her alimentary and cosmetic habits on the studied area during the study.

Exclusion Criteria:

In term of population :

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Minor subject.
4. Major subject who is under guardianship or who is not able to express her consent.
5. Subject in a social or sanitary establishment.
6. Subject suspected to be non-compliant according to the investigator's judgment.

   In term of associated pathology :
7. Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk.
8. Subject suffering from a severe or progressive disease.
9. Subject with known history of or suffering from skin disease that may interfere with evaluation of the study results and/or subject safety.
10. Subject having history of severe allergy or anaphylactic shock including known risk of hypersensitivity to one of the components of the composition of the product

    Related to previous or ongoing treatment :
11. Subject undergoing a topical treatment on the test area or a systemic treatment:

    * anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study;
    * corticosteroids during the 2 previous weeks and during the study;
    * retinoids and/or immunosuppressors during the 3 previous months and during the study;
    * any medication stabilized for less than one month.
12. Subject having started or changed her oral contraceptive or any other hormonal treatment during the three previous months.
13. Subject having done facial skin care like peeling, mask… during the previous 2 weeks and during the study.
14. Subject having used oral nutritional supplements and/or vitamin supplementation during the previous month and during the study

    In term of lifestyle :
15. Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen during the study;
16. Subject having used topical products containing actives substances during the previous 2 weeks and during the study
17. Subject planning to change her life habits during the study.
18. Subject with unstable eating habits or planning to change them during the study
19. Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 5 cigarettes per day).

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 108 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on skin translucency parameter Alpha at 84 days | From enrollment to 84 days of supplementation
  The skin translucency parameter Alpha is measured with translucency meter

SECONDARY OUTCOMES:
Change from baseline on skin translucency parameters Alpha, Area and K at 28 days and 84 days | From enrollment to 28 days of supplementation
  The skin translucency parameters Alpha, Area and Kis are measured with translucency meter
Change from baseline on skin complexion radiance at 14, 28, 56 and 84 days | From enrollment to 14, 28, 56 and 84 days of supplementation
  Skin complexion radiance measured with Colorface®
Change from baseline on pigment spot at 14, 28, 56 and 84 days | From enrollment to 14, 28, 56 and 84 days of supplementation
  Pigment spot measured with Colorface®
Change from baseline on skin firmness, elasticity and fatigability at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Skin firmness, elasticity and fatigability measured with Cutometer®
Change from baseline on Trans Epidermal Water Loss at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Trans Epidermal Water Loss measured with Tewameter®
Product safety | From enrolment to 84 days
  Safety assessed by the collection of adverse events and concomitant treatments throughout the study

OTHER OUTCOMES:
Change from baseline on skin pH at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Skin pH measured with pH meter
Change from baseline on blood flow at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Blood flow measured with Laser speckle blood flow imager®
Change from baseline on subject quality of life at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Quality of life assessed using the questionnaire SF-12 completed by the subjects
Change from baseline on subject satisfaction at 28 and 84 days | From enrollment to 28 and 84 days of supplementation
  Subject satisfaction assessed with a subjective evaluation questionnaire developed by the Sponsor completed by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Sarah ZENG, Principal Investigator — EUROFINS CONSUMER PRODUCT TESTING (Guangzhou)Co.,Ltd.
Locations (1):
- EUROFINS CONSUMER PRODUCT TESTING (Guangzhou)Co.,Ltd., Guangzhou, China

IPD SHARING:
Plan to Share IPD: No